CLINICAL TRIAL: NCT03737773
Title: Randomized Double-blind Study on the Effect of Orthoptic Rehabilitation in Pisa Syndrome Associated With Parkinson's Disease
Brief Title: Prismatic Lenses in the Pisa Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Nicola Modugno, Neurologist, Head of Parkinson Center, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDNM-01
Record Dates: First submitted 2018-10-30; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Pisa Syndrome; Parkinson' Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group prisms (Active Comparator): Patients that receive active prismatic lenses
  Interventions: Other: glasses (prismatic lenses)
- group placebo lenses (Placebo Comparator): Patients that receive non-active prismatic lenses
  Interventions: Other: glasses (neutral)

INTERVENTIONS:
Other: glasses (prismatic lenses)
  Arms: group prisms
Other: glasses (neutral)
  Arms: group placebo lenses

SUMMARY:
Non-pharmacological interventional pilot study on the effect of prismatic glasses for the improvement of Pisa syndrome in Parkinson's disease.

The study involves 40 patients, of whom 20 receive active treatment and 20 slow placebo. At the end of the study, all patients receive corrective lenses in compassionate use if the study yields positive results.

DETAILED DESCRIPTION:
In previous cases of patients with Parkinson's disease and Pisa Syndrome, the investigators found a slight improvement in the dystonia of the trunk after the application of prismatic lenses.

The current study provides the involvement of 40 patients with Parkinson's disease, of which twenty treated with permanent prismatic optical correction, and twenty treated with neutral optical correction or with the only optical correction of the refractive basic defects (placebo).

The protocol provides the collection of these data:

* Personal data (date of birth, sex, marital status, profession)
* General history (weight, height, non-neurological and neurological concomitant pathologies, medical conditions that may be associated or predisposing patients to PS, non-antiparkinsonian therapy in progress)
* Specific history for PD (year from the first diagnosis of PD, year of appearance of the first motor symptoms of PD, type and distribution of motor symptoms at the onset)
* Pharmacological history of PD (year of initiation of the first treatment for PD, which drugs (s), antiparkinsonian therapy in progress)
* Neurological Evaluation in ON: UPDRS I, II, III and IV (III: also items-20-26 right and left side), Hoehn-Yahr stage;
* Specific history for PS;
* Detection of some information about the patients' perception of having the torso tilted sideways, direction of inclination, how long it is present, how long it is manifested, conditions in which this inclination is present (standing, sitting, etc.) )
* Presence of low back pain and pain intensity measured with the Visual Analogue Scale (VAS).

Clinical and kinematic evaluation of PS:

* The amount of dystonia measured in degrees with the patient positioned against the wall against a dedicated protractor. This measurement is photographed.
* Static and dynamic kinematic evaluation (gait analysis) according to the following protocol: 30 seconds stationary in orthostatic position, shoulders to the cameras, about 5 steps forward, stationary in orthostatic position while fixing visual stimulation points placed on the wall, 30 second stationary in an orthostatic position after having covered a section of the corridor in front of the kinematic evaluation room.

Orthoptic evaluation:

complete orthoptic evaluation and prescription of personalized prismatic lenses, randomizing the patient on active or slow-moving placebo lenses with respect to the other experimenters and the patient.

Flowchart of visits:

Screening: the neurologist selects the patient according to the eligibility criteria indicated above and verifies the patient's willingness to participate.

Randomization: the patient undergoes clinical and kinematics evaluation of the PS, orthoptic examination and randomization on active lenses and placebo.

Study times:

T0: randomization and prescription of lenses T1: check after 1 month from the use of lenses

Patients are recruited at the Parkinson's Center of the IRCCS Neuromed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Diagnosis of PD according to the diagnostic criteria of the United Kingdom Brain Bank with or without dementia (but with MMSE> 14)
* Hoehn-Yahr Stadium from 1 to 4
* Signature of Informed Consent and the privacy form

Exclusion Criteria:

* Patients with morphostructural changes in the spine that exclude the diagnosis of PS.
* Patients with symptoms and signs compatible with atypical parkinsonism
* Patients affecd by PD treated with antagonist drugs for central dopaminergic receptors (first generation antipsychotics and second generation with the exception of clozapine and quetiapine, antiemetic, prokinetic, etc.) in the last 6 months before enrollment
* Patients with a history of major spinal surgery (tumors, infections, ankylosing spondylitis, paraneoplastic syndromes)
* Other neurological diseases.
* Patients with manifested disorders of eeye movement disorders prior to the diagnosis of PD
* Patents with abnormalities of normal binocular vision
* Patients with amblyopia, medium or high anisometropy,
* Patients with a binocular vision acuity less than 7/10
* Patients with evolved cataracts
* Pateints with glaucoma
* Patients with active maculopathies
* Patients with severe mono or binocular visual field depressions of different origins Patients with astigmatisms higher than 3 dioptres, hypermetropias or myopias greater than 3 dioptres

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Determine the change of dystonia in Pisa syndrome with the use of prisms | 1 month
  Verify the possible variation of dystonia in patients affected by Pisa Syndrome after the use for a month of prismatic lenses prescribed during the randomization phase with the aid of a wall protractor through the recording of the amount of dystonia measured in degrees with the patient positioned against the wall against a dedicated protractor. This measurement is photographed.
Determine the kinematic variation in Pisa Syndrome with the use of prisms | 1 month
  Verify the static and dynamic kinematic variation in patients affected by Pisa Syndrome after the use for a month of prismatic lenses prescribed during the randomization phase and according to the following protocol: 30 seconds stationary in orthostatic position, shoulders to the cameras, about 5 steps forward, stationary in orthostatic position while fixing visual stimulation points placed on the wall, 30 second stationary in an orthostatic position after having covered a section of the corridor in front of the kinematic evaluation room.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Modugno, MD, PHD, Principal Investigator — Neuromed IRCCS

IPD SHARING:
Plan to Share IPD: No